CLINICAL TRIAL: NCT05770830
Title: Correlation Between Esophageal Temperature and Skin Temperature Measured by 3M™ Bair Hugger™ in Trauma Patients
Brief Title: Correlation Between Esophageal Temperature and Skin Temperature in Trauma Patients
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, Assistana professor, Ajou University School of Medicine
Other Study IDs: AJOUIRB-MDB-2021-557
Record Dates: First submitted 2023-03-04; First posted 2023-03-16 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Core Temperature; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Esophageal temperature: Esophageal temperature
  Interventions: Device: Esophageal temperature
- Skin core temperature: Skin core temperature
  Interventions: Device: Skin core temperature

INTERVENTIONS:
Device: Esophageal temperature — Temperature data measured by esophageal temperature probe (disposable probe, Ace-medical, Seoul, Korea)
  Groups: Esophageal temperature
Device: Skin core temperature — Temperature data measured by skin core temperature device measured by 3M™ Bair Hugger™
  Groups: Skin core temperature

SUMMARY:
The goal of this retrospective data-based study is to investigate the correlation between esophageal temperature and skin core temperature in trauma patients who underwent emergency surgery.

Based on the medical records of patients who applied both temperature measurements simultaneously, the correlation between the skin core temperature and the esophageal temperature was investigated

DETAILED DESCRIPTION:
Hypothermia is known to be one of the factors that increase mortality rate in trauma patients. Therefore it is important to measure and manage the core temperature in trauma patients.

Esophageal temperature is common method to measure core temperature in patients undergoing surgery under general anesthesia. However, it is not applicable in patients who have not been intubated or in patients with suspected esophageal damage. In addition, esophageal temperature probe is twisted in the mouth and does not reflect core temperature properly.

3M™ Bair Hugger™ temperature monitoring system was developed to measure the core temperature by attaching to the skin using zero heat flow mechanism. It is simple to apply, and available at the trauma scene.

Previous studies have reported that skin core temperature reflects core temperature well, but no studies have been conducted on trauma patients with rapid changes in the core temperature and poor perfusion state.

This retrospective data-based study investigate the medical records of trauma patients who underwent emergency surgery. Patients who applied two temperature measurements at the same time were targeted. Since this center has the system that automatically transfer the hemodynamic data of the monitor to the anesthesia record, the investigators use the anesthesia records.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients who underwent emergency surgery from January 1, 2021 to October 31, 2021
* Who applied both a esophageal thermometer and a 3M™ Bair Hugger™ temperature monitoring system at the same time

Exclusion Criteria:

* When more than half of the data is missing

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Trauma patients who underwent emergency surgery from January 1, 2021 to October 31, 2021
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
accuracy | 3 hours
  Mean difference between the two temperatures

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
We can shre the data when there is a reasonable request to the corresponding author.